CLINICAL TRIAL: NCT01207648
Title: Retrospective Cohort Study of Rebif® Use in Pediatric MS Patients
Brief Title: Retrospective Cohort Study of Rebif® Use in Pediatric Multiple Sclerosis (MS) Subjects (REPLAY)
Acronym: REPLAY
Status: Completed | Type: Observational
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR 200136-024
Record Dates: First submitted 2010-09-21; First posted 2010-09-23 (Estimated); Results first posted 2013-05-30 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-04

CONDITIONS: Multiple Sclerosis
Keywords: Interferon beta 1a; Autoimmune Diseases; Demyelinating Diseases; Immune System Diseases; Immunologic Factors; Nervous System Diseases; Physiological Effects of Drugs; Demyelinating Autoimmune Diseases, CNS; Autoimmune Diseases of the Nervous System; Retrospective Cohort Study
MeSH Terms: conditions — Multiple Sclerosis; Autoimmune Diseases; Demyelinating Diseases; Immune System Diseases; Nervous System Diseases; Demyelinating Autoimmune Diseases, CNS; Autoimmune Diseases of the Nervous System | interventions — Interferon beta-1a

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Retrospective Cohort: Pediatric participants including both children (aged less than 12 years) and adolescents (aged 12 to less than 18 years) who were exposed to Rebif® for treatment of demyelinating events were observed in this retrospective cohort study. In this study, medical records of participants evaluated between 1997 to 2009 were reviewed. The observation period started with the first medical record available on site till last medical record available on site or the end of the observation period (31 December 2009), whichever occurred first.
  Interventions: Drug: Rebif®

INTERVENTIONS:
Drug: Rebif® — This is an retrospective cohort study in Pediatric participants including both children (aged less than 12 years) and adolescents (aged 12 to less than 18 years) who were exposed to Rebif® for treatment of demyelinating events (Dose regimen as per investigator's decision)

SUMMARY:
The aim of this retrospective study is to review and describe safety, tolerability and efficacy of Rebif® (subcutaneous interferon [IFN]-beta-1a) in children and adolescents, using information already recorded in medical records. The study duration is 13 July 2010 (first data collected) to 13 July 2011 (last data collected). In this study, Data of the subjects evaluated between 1997 and 2009 was observed.

ELIGIBILITY:
Inclusion Criteria:

* Received one or more injections of Rebif® for treatment of a demyelinating event
* Be younger than 18 years of age at time of Rebif® treatment initiation
* Rebif® therapy must have been initiated before June 30, 2009

Exclusion Criteria:

No exclusion criteria are applied

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Every eligible subject at participating centers: subjects who have received one or more injections of Rebif® for treatment of a demyelinating event before the age of 18 and before the 30th June 2009.
Sampling Method: Non-Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2010-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Inc., a subsidiary of Merck KGaA, Darmstadt, Germany
Locations (18):
- United States (6):
  - Research Site, Birmingham, Alabama
  - Research Site, San Francisco, California
  - Research Site, Boston, Massachusetts
  - Research Site, Buffalo, New York
  - Research Site, Rochester, New York
  - Research Site, Stoney Brook, New York
- Research Site, Buenos Aires, Argentina
- Research Site, Toronto, Canada
- Research Site, Le Kremlin-Bicêtre, France
- Italy (6):
  - Research Site, Bari
  - Research Site, Catania
  - Research Site, Gallarate
  - Research Site, Milan
  - Research Site, Rome
  - Research Site, Torino
- Research Site, Moscow, Russia
- Research Site, Tunis, Tunisia
- Research Site, Maracaibo, Venezuela

RESULTS

PARTICIPANT FLOW:
Groups:
- Retrospective Cohort: Pediatric participants including both children (aged less than 12 years) and adolescents (aged 12 to less than 18 years) who were exposed to Rebif® for treatment of demyelinating events were observed in this retrospective cohort study. In this study, medical records of participants evaluated between 1997 to 2009 were reviewed. The observation period started with the first medical record available till last medical record available on site or the end of the observation period (31 December 2009), whichever occurred first.
Period: Overall Study
Arm/Group | Retrospective Cohort
Started | 307
Completed | 307
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Retrospective Cohort
Number analyzed (Participants) | 307
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.0 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 190
  Male | 117

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Pre-specified Medical Events
Description: These pre-specified medical events categories were evaluated: injections site reactions, flu-like symptoms, hepatic disorders, blood cell disorders, allergic reactions, epilepsy and convulsive disorders, thyroid dysfunction, autoimmune diseases, bone/epiphyseal and cartilage disorders, serious infections, malignancies. Each category defined by group of events which best fit the medical concept either using a standard medical dictionary for regulatory activities (MedDRA) Query (SMQ) e.g., Malignancies was defined by the SMQ Malignancies (narrow scope) containing more than 1800 different preferred terms (PTs) (including procedures and lab tests) or using a customized query, e.g., Serious infections was defined by all PTs assessed as serious in System Organ Class (SOC) Infections and Infestation. Participants may be represented in more than once in a category (Participants could have reported several medicals events pertaining to a specific category) as well as in more than one category.
Time Frame: Start of observation period (first medical record available on site) up to last medical record available on site or the end of the observation period (31 December 2009), whichever occurred first.
Population: Total analysis set included all the participants who were exposed to Rebif® for treatment of demyelinating event and were evaluated in this retrospective study.
Measure: Number; unit: Participants
Arm/Group | Retrospective Cohort
Number analyzed (Participants) | 307
Participants
  Injections site reactions | 85
  Flu-like symptoms | 75
  Hepatic disorders | 44
  Blood cell disorders | 14
  Allergic reactions | 5
  Epilepsy and convulsive disorders | 5
  Thyroid dysfunction | 3
  Autoimmune diseases | 2
  Bone/epiphyseal and cartilage disorders | 2
  Serious infections | 2
  Malignancies | 1

2. Primary Outcome: Number of Participants With Serious Medical Events, and Non-serious Medical Events (Reported by the Investigator as Related to Rebif®)
Description: Medical events in the retrospective study are equivalent to adverse events in a prospective clinical study. A medical event was defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to baseline during a clinical study with an investigational medicinal product (IMP), regardless of causal relationship and even if no IMP has been administered. Serious medical event: A medical event that resulted in death; was life threatening; resulted in persistent/significant disability/incapacity; resulted in/prolonged an existing in-patient hospitalization; was a congenital anomaly/birth defect; or was a medically important condition. Participants may be represented in more than one category as participant who had experienced serious medical event may also had experienced non-serious medical event reported by the Investigator as related to Rebif®, so in that case it will be counted in both the categories.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Retrospective Cohort
Number analyzed (Participants) | 307
Participants
  Serious medical events | 12
  Non-serious medical events | 184

3. Primary Outcome: Number of Participants With Abnormal Laboratory Parameters
Description: Laboratory parameters assessed for abnormality were: total white blood cell count (Neutrophils, Lymphocytes, Leukocytes, Monocytes, Eosinophils and Basophils), differential hematogram (Hematocrit, Erythrocytes, Hemoglobin, and Platelet), aspartate aminotransferase (AST), alanine aminotransferase (ALT), and thyroid tests (including Triiodothyronine, Thyroxine, Thyroperoxidase Antibody and Thyroid-Stimulating Hormone). Due to the retrospective nature of the study, laboratory data should be interpreted with caution as data were not collected according to a specific time schedule and the time on study per participant was not standardized.
Time Frame: as for outcome 1
Population: Total analysis set included all the participants who were exposed to Rebif® for treatment of demyelinating event and were evaluated in this retrospective study. 'n' signifies number of participants who were evaluable for the specified categories.
Measure: Number; unit: Participants
Arm/Group | Retrospective Cohort
Number analyzed (Participants) | 307
Participants
  Alanine Aminotransferase (n=195) | 74
  Aspartate Aminotransferase (n=194) | 59
  Basophils (n=190) | 4
  Eosinophils (n=190) | 13
  Erythrocytes (n=193) | 28
  Hematocrit (n=196) | 38
  Hemoglobin (n=196) | 33
  Leukocytes (n=200) | 45
  Lymphocytes (n=190) | 55
  Monocytes (n=189) | 18
  Neutrophils (n=192) | 46
  Platelet (n=196) | 13
  Thyroid-Stimulating Hormone (n=116) | 4
  Thyroperoxidase Antibody (n=71) | 2
  Thyroxine (n=99) | 3
  Triiodothyronine (n=80) | 4

4. Secondary Outcome: Annualized Medically Confirmed Clinical Relapses Rate Prior to Rebif® Initiation and During Rebif® Treatment
Description: Medically confirmed clinical relapses were defined as the emergence of new neurological symptoms that occurred more than 30 days after a previous attack and persisted for more than or equal to 24 hours in the absence of known inter-current illness. Annualized relapse rate was defined as number of attacks per year.
Time Frame: as for outcome 1
Population: Multiple sclerosis (MS) analysis set is a subset of the "Retrospective Cohort" set included all participants with a final diagnosis of MS. 'N' (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Number; unit: Attacks per year
Arm/Group | Retrospective Cohort
Number analyzed (Participants) | 298
Attacks per year
  Prior to Rebif® initiation | 1.79
  During Rebif® treatment | 0.47

5. Secondary Outcome: Time to First Medically Confirmed Clinical Relapse Post-Rebif® Initiation
Description: Medically confirmed clinical relapses were defined as the emergence of new neurological symptoms that occurred more than 30 days after a previous attack and persisted for more than or equal to 24 hours in the absence of known inter-current illness.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Retrospective Cohort
Number analyzed (Participants) | 298
Months | 19.5 [14.5 to 27.2]

ADVERSE EVENTS:
Time Frame: Start of observation period (first medical record available on site) up to last medical record available on site or the end of the observation period (31 December 2009), whichever occurred first.
Description: A medical event was defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to baseline during a clinical study with an IMP, regardless of causal relationship and even if no IMP has been administered.
Arm/Group | Retrospective Cohort
Serious Adverse Events (participants affected / at risk) | 12/307
Other Adverse Events (participants affected / at risk) | 184/307
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Retrospective Cohort (N=307)
Injection site injury (General disorders) | 1
Injection site necrosis (General disorders) | 1
Irritability (General disorders) | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Cellulitis (Infections and infestations) | 1
Injection site cellulitis (Infections and infestations) | 1
Convulsion (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Hallucination, auditory (Psychiatric disorders) | 1
Suicidal behaviour (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Liver function test abnormal (Investigations) | 1
Appendicectomy (Surgical and medical procedures) | 1
Omentectomy (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Retrospective Cohort (N=307)
Influenza like illness (General disorders) | 75
Injection site erythema (General disorders) | 48
Injection site pain (General disorders) | 34
Pyrexia (General disorders) | 9
Fatigue (General disorders) | 5
Chills (General disorders) | 4
Injection site haematoma (General disorders) | 4
Injection site reaction (General disorders) | 4
Alanine aminotransferase increased (Investigations) | 13
Hepatic enzyme increased (Investigations) | 9
Liver function test abnormal (Investigations) | 8
Aspartate aminotransferase increased (Investigations) | 7
Headache (Nervous system disorders) | 19
Leukopenia (Blood and lymphatic system disorders) | 7
Liver disorder (Hepatobiliary disorders) | 7
Nausea (Gastrointestinal disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 4
Depression (Psychiatric disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other